CLINICAL TRIAL: NCT01085448
Title: Identifying the Subgroup of Patient With Mechanical Low Back Pain Who Have Clinical Lumbar Instability
Brief Title: Clinical Prediction Rule for Clinical Lumbar Instability
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of timely recruitment of subjects
Sponsor: Drexel University (Other)
Responsible Party: Principal Investigator, Sheri Silfies, Associate Professor, Drexel University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DRX18590
Record Dates: First submitted 2010-03-10; First posted 2010-03-11 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2013-11

CONDITIONS: Low Back Pain
Keywords: low back pain; core stabilization; physical therapy
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Low back pain (Other): Individuals with current low back pain.
  Interventions: Other: Core Stabilization

INTERVENTIONS:
Other: Core Stabilization — The 8-week program emphasizes use of specific local stabilizing muscles (transverse abdominis[TrA], lumbar multifidus[LM]) to restore active control to the trunk. Emphasis is on training isometric co-contractions and a progression (3 stages) based upon a motor learning paradigm.
  Stage 1: neutral position of the spine and activation of the TrA and LM. Performance feedback is emphasized and monitored through observation and palpation.
  Stage 2: maintenance the co-contraction while performing movements of the trunk and the upper and lower extremities. Trunk conditioning is also emphasized. Feedback is gradually reduced.
  Stage 3: maintenance of the co-contraction while performing exercises on an unstable surface or during perturbation of the activity. Random practice patterns are used to enhance motor learning.

SUMMARY:
The aim of this study is to determine if assessment of additional measures of trunk neuromuscular control will improve the ability to identify patients with low back pain who successfully respond to trunk stabilization exercises.

Question: What clinical characteristics are associated with patients that respond positively to a program of core stabilization exercises?

Hypothesis: Clinical characteristics that show a decrease in trunk motor control will be associated with a positive response to stabilization exercises.

DETAILED DESCRIPTION:
Clinical identification of individuals with mechanical low back pain who would benefit from a program of stabilization exercises has been a struggle for the physical therapy profession. While changes in trunk muscle recruitment and motor control have been linked to patients with chronic low back pain and hypothesized to be adaptations for spinal instability, this has not been systematically established. However, a connection between spinal instability, poor trunk motor control, and low back pain is plausible. The real problem lies with the clinical identification of the subgroup of patients in either the acute or chronic phases of low back dysfunction who would most benefit from this approach to intervention.

In creating their preliminary clinical prediction rule, Hicks et al (2005), looked at many variables including patient demographics and characteristics, hip and trunk motion, special tests for instability, and functional measures of muscle performance. However, measures of the performance of core stabilizing muscles and assessment of trunk dynamic control/ coordination were not included as potential variables. The aim of this study is to determine if assessment of additional measures of trunk neuromuscular control will improve the ability to identify patients with low back pain who successfully respond to trunk stabilization exercises.

ELIGIBILITY:
Inclusion Criteria:

1. duration of the current episode of low back pain less than 3 months,
2. average pain intensity over past 3 days at least 4 on an 11 point (0 = no pain, 10 = worst pain ever) numeric pain rating scale,
3. no medical intervention for low back pain in last 6 months,
4. Oswestry score greater than 25%

Exclusion Criteria:

1. permanent structural spinal deformity (e.g., scoliosis)
2. history of spinal fracture or diagnosis of osteoporosis
3. diagnosis of inflammatory joint disease
4. signs of systemic illness or suspected non-mechanical LBP (i.e. spinal tumor or infection)
5. previous spinal surgery
6. frank neurological loss, i.e., weakness and sensory loss
7. history of neurologic disease that required hospitalization,
8. active treatment of another medical illness that would preclude participation in any aspect of the study or any lower extremity injury that would potentially alter trunk movement in standing
9. leg length discrepancy of greater than 2.5 cm.
10. pregnancy
11. vestibular dysfunction

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-03; Primary Completion 2012-08 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index | Baseline, 8 weeks
  measure of functional limitation

SECONDARY OUTCOMES:
Numeric Pain Scale | Baseline, 8 weeks
  measure of preceived pain

CONTACTS AND LOCATIONS:
Overall Officials: Sheri P. Silfies, PT, PhD, Principal Investigator — Drexel University
Locations (2):
- United States (2):
  - Drexel University, Philadelphia, Pennsylvania
  - Optimum Physical Therapy Associates, West Chester, Pennsylvania